CLINICAL TRIAL: NCT02894372
Title: Faringomoss Effectiveness in Inhibiting Acute Throat Pain and Discomfort
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lithuanian University of Health Sciences (Other)
Collaborators: Klaipėda University (Other); Vita Longa Clinic (Unknown)
Responsible Party: Principal Investigator, Nora Siupsinskiene, Professor, Doctor of Medicine and Doctor of Philosophy (PhD), Lithuanian University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Far1
Record Dates: First submitted 2016-06-19; First posted 2016-09-09 (Estimated); Last update posted 2017-03-13 (Actual); Status verified 2017-03

CONDITIONS: Spraying Behavior; Mouth Diseases; Throat Diseases; Throat Pain
Keywords: Oral spray; Topical sprays; Faringomoss; Local phytotherapy
MeSH Terms: conditions — Mouth Diseases; Pharyngitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Subjects with oral spray 1 (Experimental): Research subjects, who got oral spray 1. Spray was used 3 times a day 3 sprays a time for seven days. Spray 1 was Faringomoss or simple oily oral spray (unknown because of double blind method).
  Interventions: Device: Oral spray 1
- Subjects with oral spray 2 (Experimental): Research subjects, who got oral spray 2. Spray was used 3 times a day 3 sprays a time for seven days. Spray 2 was Faringomoss or simple oily oral spray (unknown because of double blind method).
  Interventions: Device: Oral spray 2

INTERVENTIONS:
Device: Oral spray 1 — Research participants got topical oral spray immediately after surgery (hospital patients) and from the first doctor visit with pharyngeal disease (clinic outpatients).
  Arms: Subjects with oral spray 1
Device: Oral spray 2 — Research participants got topical oral spray immediately after surgery (hospital patients) and from the first doctor visit with pharyngeal disease (clinic outpatients).
  Arms: Subjects with oral spray 2

SUMMARY:
The purpose of the study was to assess the effectiveness of Faringomoss in reducing the throat discomfort and pain in patients with acute throat diseases and postoperative patients after throat surgeries.

DETAILED DESCRIPTION:
Study objectives were:

1. To asses the symptoms of throat pain and discomfort after pharyngeal surgery in early postoperative period.
2. To evaluate those symptoms also in outpatient subjects with acute throat pain and discomfort.
3. To compare the data of different groups of patients who had received the topical throat spray with the placebo group.
4. To estimate the gender, age and surgery impact on the results.
5. To record the side effects of the topical sprays.

Patients were selected from Lithuanian University of Health Sciences Ear-Nose-Throat department and Vita Longa Clinic outpatients.

In random order research participants got a topical spray to use for 7 days after the surgery or from the start of acute throat infection. Neither the patient nor the investigator did not know if it was the medical device (Faringomoss) or the placebo. All the participants got a standard care and treatment with non-steroidal anti-inflammatory drugs.

The intent was to investigate about 70 - 80 subjects.

All the research subjects were tested using objective methods.

The confidentiality of the participation was guaranteed. The names were anonymous. The results were summarized.

Faringomoss is a topical spray, approved as a medical device. It is not harmful because it is made of vegetable oils.

ELIGIBILITY:
Inclusion Criteria:

* Patients after throat surgeries: tonsillectomy, adenotonsillectomy, uvulopalatoplasty, uvulopalatopharyngoplasty
* Patients with acute throat diseases: pharyngitis, tonsillitis, pharyngotonsillitis

Exclusion Criteria:

* Purulent infection
* Refusal to participate
* Allergy to tested material

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2015-01; Primary Completion 2016-11-01 (Actual); Study Completion 2016-12-30 (Actual)

PRIMARY OUTCOMES:
Symptoms changes during treatment assessed using the 100 mm visual analog scale (VAS) | The first, third, fifth and seventh treatment days
  Scale assessment: 0 point - no symptom, 100 points - strong symptom manifestation. Evaluated symptoms are: throat pain, ear pain, swallowing pain, difficult mouth opening, difficult swallowing, impaired nutrition, general condition, how symptoms are effecting life. If additional symptoms occur during investigation period, they are assessed too.

SECONDARY OUTCOMES:
Pharyngoscopic examination of the oropharyngeal mucosa of throat using Likert scale | After 7 days of treatment
  Mucosal erythema, swelling, erosion, fibrin plaque, fistulas are evaluated using three points (0-2) Likert scale.
Secondary bleeding after surgery | Up to 7 days
  We note if there was a bleeding after throat surgery during investigation time.
Use of medicines | Up to 7 days
  We evaluate the amount of used standardized analgesics/anti-inflammatory drugs.
Period of time to notice the effect | Up to 7 days
  We measure how many days or hours it took for the patient to notice the effect of the medical device.

CONTACTS AND LOCATIONS:
Overall Officials: Nora Siupsinskiene, Professor, Principal Investigator — Hospital of Lithuanian University of Health Sciences, Otorhinolaryngology department; Nora Siupsinskiene, Professor, Principal Investigator — Klaipėda University
Locations (1):
- Lithuanian University of Health Sciences, Kaunas, Lithuania

IPD SHARING:
Plan to Share IPD: Undecided